CLINICAL TRIAL: NCT04605146
Title: Impact of Telemonitoring for the Management of Side Effects in Patients with Melanoma, Lung or Renal Cancer, Treated with Immunotherapy Combination of Nivolumab and Ipilimumab or Adjuvant Nivolumab Monotherapy
Acronym: MONITOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL20_0492; 2020-A02372-37 (Other: ID-RCB)
Record Dates: First submitted 2020-10-16; First posted 2020-10-27 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Melanoma; Lung Cancer; Renal Cancer
Keywords: Tele-monitoring; nivolumab; ipilimumab; immunotherapy
MeSH Terms: conditions — Melanoma; Lung Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tele-monitoring group (Experimental): In the experimental group, in addition to routine practice, each patient will benefit of a tele-monitoring of one year, and a long term follow-up up to 5 years to evaluate the Overall Survival and the Progression-Free Survival. Quality of life questionnaire will also be filled in at inclusion, M3 and M12.
  50 patients are expected in this arm.
  Interventions: Behavioral: Tele-monitoring
- Control group (No Intervention): In the control group, patients will have a routine follow-up as per institutional practice, and a long term follow-up up to 5 years to evaluate the Overall Survival and the Progression-Free Survival. Quality of life questionnaire will also be filled in at inclusion, M3 and M12.
  50 patients are expected in this arm.

INTERVENTIONS:
Behavioral: Tele-monitoring — The tele-monitoring will consist in filling in a specific questionnaire once a week in the first 6 months, every 2 weeks until 12 months, and on-demand (in case of upcoming toxicity, at any time). These questionnaires will be reviewed by a coordinating nurse. According to the result of the questionnaire, the coordinating nurse will adapt patients' management, either by giving them a phone call, or inviting them to directly contact their medical department, or even plan an emergency hospitalization if necessary. The coordinating nurse will closely work with the investigator to adapt patients' management.
  Quality of life questionnaire (FACT-G) will also be filled in at inclusion, M3 and M12.
  Arms: Tele-monitoring group

SUMMARY:
The ipilimumab and nivolumab combination is now part of the standard of care for the treatment of melanoma, renal and lung cancer patients. Grade 3/4 adverse events (AEs) occur in 30 to 60% of patients included in clinical trials. Grade 3/4 AEs are more frequently observed (50-60% of patients) in melanoma because ipilimumab is administrated at 3mg/kg in this population. Among these AEs, early detection of immune related AEs is critical to an adequate medical management. In this context, dedicated tools for remote monitoring of these patients are crucial.

The investigators developed within the Immucare consortium a simplified medical questionnaire which is addressed weekly to the patients. This questionnaire along with an algorithm gives to the clinician regular feedback on their patients' general symptoms. The investigators herein want to evaluate in a randomized prospective trial the efficacy of this remote monitoring to reduce the time between the start of AE and the reporting to the medical team, which could lead to detect and treat earlier AEs induced by nivolumab and ipilimumab in the melanoma, lung and renal cancer patients' population.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients diagnosed with melanoma, or lung cancer or renal cancer
* Patients starting a treatment with a combination of immunotherapy of nivolumab + ipilimumab (NB: patients who have already received immunotherapy in the past may be included)
* Patients comfortable with the use of digital tools and computing
* Patients who agree to participate to the telemonitoring and signed consent form

Exclusion Criteria:

* Pregnant, parturient and lactating women
* Patients under legal protection measure or deprived of their liberty
* Patients not affiliated to a social security scheme (schemes such as the AME) or beneficiaries of a similar regime (foreign person, outside the EU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2028-11-05 (Estimated); Study Completion 2028-11-05 (Estimated)

PRIMARY OUTCOMES:
Delay between the start of a side effect and reporting to the medical team (average number of days per patient). | 12 months
  The delay between the start of a side effect and medical information will be calculated for each AE and average per patient in each of the two groups studied, with its 95% confidence interval.The delays of the two groups will be compared using a Mann-Whitney test.

SECONDARY OUTCOMES:
Levels of morbidity based on CTC-AE v5 (all toxicities) | 12 months
  Levels of morbidity based on CTC-AE v5 (all toxicities) will be compare using a generalised log linear regression. In case of several AEs, the average medical information per patient will be considered.
Number of treatment interruptions and number of days of treatment delays interruptions, number of treatment discontinuation, number of dose reductions and and percentage of dose reduction | 12 months
  Number of treatment interruptions and number of days of treatment delays interruptions, number of treatment discontinuation, number of dose reductions and and percentage of dose reduction will be compared in the two groups using a Mann-Whitney test
Number of admissions in the emergency room | 12 months
  Number of admissions in the emergency room will be compared in the two groups with a Wilcoxon rank sum test. The rate of admissions per patient-years will be calculated and compared between the 2 groups with a Negative Binomial generalized linear regression model accounting for overdispersed data and correlated events, using the log of follow-up time as an offset.
Number of unplanned hospitalizations | 12 months
  Number of unplanned hospitalizations will be compared in the two groups with a Wilcoxon rank sum test.
  The hospitalizations per patient-years will be calculated and compared between the 2 groups with a Negative Binomial generalized linear regression model accounting for overdispersed data and correlated events, using the log of follow-up time as an offset.
Number of contact with general practitioner | 12 months
  Number of contact with general practitioner will be compared in the two groups with a Wilcoxon rank sum test.
benefit for clinicians: interview of clinicians on their opinion on the self-monitoring, evaluation to the impact on the consultations during the first year of treatment, assessed with satisfaction questionnaires | Month 12
  benefit for clinicians will be compared in the 2 groups with adequate test according to the retained satisfaction scale
Number of AE identified by clinicians | 12 months
  Number of AE identified by clinicians will be compared in the two groups with a Wilcoxon rank sum test.
  In addition, the competitive risk of death with the recurrent events process will be explored using a joint frailty model (Rondeau V. et al. Joint frailty models for recurring events and death using maximum penalized likelihood estimation: application on cancer events. Biostatistics (2007), 8, 4, pp. 708-721).
Overall quality of Life assessed with standardized QoL questionnaires (FACT-G) | 12 months
  Overall quality of Life will be described and compared between the two groups with the Student t-test, or the Wilcoxon rank-sum test in case of non-normality of the distributions. All data recorded at the follow-up visits will be considered, whatever the actual date of the visit
Adherence: The number of full symptoms report completions and adherence to the completion schedule | 12 months
  Adherence will be described in the experimental group. All data recorded at the follow-up visits will be considered, whatever the actual date of the visit.

OTHER OUTCOMES:
Overall Survival and Progression Free Survival assessed at 1 year after inclusion | At 1 year after inclusion
  Overall Survival and Progression Free Survival will be estimated based on computed time between randomisation and date of the first event which ever would it be (death or progression) or date of last follow-up. Survival probabilities will be estimated suing Kaplan Meier approach
Overall Survival and Progression Free Survival assessed at 2 years after inclusion | At 2 years after inclusion
  Overall Survival and Progression Free Survival will be estimated based on computed time between randomisation and date of the first event which ever would it be (death or progression) or date of last follow-up. Survival probabilities will be estimated suing Kaplan Meier approach
Overall Survival and Progression Free Survival assessed at 5 years after inclusion | At 5 years after inclusion
  Overall Survival and Progression Free Survival will be estimated based on computed time between randomisation and date of the first event which ever would it be (death or progression) or date of last follow-up. Survival probabilities will be estimated suing Kaplan Meier approach

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane DALLE, Principal Investigator — Department of Dermatology, HCL-Cancer Institute
Locations (10):
- France (10):
  - Groupement hospitalier Est - Multidisciplinary oncological platform, Bron
  - Hôpital Louis Pradel - Department of Pneumology, Bron
  - University hospital of Grenoble Alpes - Department of dermatology, Grenoble
  - University hospital of Grenoble Alpes - Department of Medical Oncology, Grenoble
  - Hôpital de la Croix Rousse - Department of Pneumology, Lyon
  - Hôpital Edouard Herriot - Department of urology, Lyon
  - Centre Hospitalier Lyon Sud - Department of Medical Oncology, Pierre-Bénite
  - Hôpital Lyon Sud - Department of Dermatology, HCL-Cancer Institute, Pierre-Bénite
  - Hôpital Lyon Sud - Department of pneumology,Thoracic oncology, Pierre-Bénite
  - University hospital of Saint-Etienne - Department of dermatology, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.chu-lyon.fr/fr/cancer-immucare